CLINICAL TRIAL: NCT04453137
Title: Multicenter, Double-Blind, Randomized, Parallel-group, Study Evaluating PK, Efficacy, Safety, and Immunogenicity in Patients With Plaque Psoriasis Receiving Humira® or AVT02 Followed by a Safety Extension Phase of AVT02
Brief Title: Pharmacokinetic, Efficacy, Safety, and Immunogenicity of AVT02 With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AVT02-GL-302
Record Dates: First submitted 2020-05-15; First posted 2020-07-01 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Adalimumab; adalimumab biosimilar HS016

STUDY DESIGN:
Intervention Model Description: Open label lead-in phase, followed by blinded 1:1 randomization with open label extension phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Humira 40 mg/mL (Adalimumab Originator) (Active Comparator): During the LeadIn Period, patients will receive Humira (initial dose of 80 mg [2 × 40 mg] administered subcutaneously [SC], followed by 40 mg SC given every other week starting 1 week after the initial dose). At Week 12, responsive patients (Psoriasis Area and Severity Index [PASI] ≥ 75 [PASI75]) will be randomly assigned in a 1:1 ratio to either of the following groups for participation in the Double-Blind Switching Module.
  Interventions: Biological: Adalimumab originator
- IC - Humira 40 mg/mL (Adalimumab Originator) (Active Comparator): patients continue to receive Humira 40 mg every other week from Week 12 until Week 26 (8 injections)
  Interventions: Biological: Adalimumab originator
- IC - Humira/AVT02 40 mg/mL (Adalimimab Biosimilar) (Experimental): patients undergo repeated switches (Sw) of AVT02 and Humira from Week 12 until Week 26:
  * Sw1-AVT02 (40 mg every other week) for 4 weeks (2 injections),
  * Sw2-Humira (40 mg every other week) for 4 weeks (2 injections),
  * Sw3-AVT02 (40 mg every other week) for 8 weeks (4 injections).
  Interventions: Biological: Adalimumab originator; Biological: Adalimumab biosimilar
- AVT02 40 mg/mL (Adalimimab Biosimilar) (Experimental): At Week 28, after the EoS IC visit, responsive patients (PASI ≥ 50 [PASI50]) will be offered to continue with the optional open-label Extension Phase (Weeks 28 to 52). AVT02 40 mg will be administered every other week starting from Week 28 (after completing EoS IC assessments), ending with the final study drug administration at Week 50. The EoS visit is planned for Week 52.
  Interventions: Biological: Adalimumab biosimilar

INTERVENTIONS:
Biological: Adalimumab originator — Subcutaneous injection every other week
  Other Names: Humira
  Arms: Humira 40 mg/mL (Adalimumab Originator); IC - Humira 40 mg/mL (Adalimumab Originator); IC - Humira/AVT02 40 mg/mL (Adalimimab Biosimilar)
Biological: Adalimumab biosimilar — Subcutaneous injection every other week
  Other Names: AVT02
  Arms: AVT02 40 mg/mL (Adalimimab Biosimilar); IC - Humira/AVT02 40 mg/mL (Adalimimab Biosimilar)

SUMMARY:
Pharmacokinetic, Efficacy, Safety, and Immunogenicity Between Patients with Moderate to Severe Chronic Plaque Psoriasis Receiving Humira® and Patients with Moderate to Severe Chronic Plaque Psoriasis

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-group study to evaluate PK, efficacy, safety, and immunogenicity between patients with moderate to severe chronic plaque psoriasis receiving Humira and patients with moderate to severe chronic plaque psoriasis undergoing repeated switches between Humira and AVT02, followed by an optional safety Extension Phase.

AVT02-GL-302 study is composed of 3 parts:

LeadIn Period: Week 1-12 - OpenLabel Treatment Switching Module: Week 12-28 - DoubleBlind Treatment Optional Extension Phase: Week 28-52 - OpenLabel Treatment

Lead-In Period:

After successfully completing Screening activities, patients will be enrolled in the LeadIn Period.

During the LeadIn Period, patients will receive Humira (initial dose of 80 mg [2 × 40 mg] administered subcutaneously [SC], followed by 40 mg SC given every other week starting 1 week after the initial dose). At Week 12, responsive patients (Psoriasis Area and Severity Index [PASI] ≥ 75 [PASI75]) will be randomly assigned in a 1:1 ratio to either of the following groups for participation in the Double-Blind Switching Module.

Switching Module:

Group 1: patients undergo repeated switches (Sw) of AVT02 and Humira from Week 12 until Week 26:

Sw1-AVT02 (40 mg every other week) for 4 weeks (2 injections), Sw2-Humira (40 mg every other week) for 4 weeks (2 injections), Sw3-AVT02 (40 mg every other week) for 8 weeks (4 injections). Group 2: patients continue to receive Humira 40 mg every other week from Week 12 until Week 26 (8 injections) The last study treatment administration in the Double-Blind Switching Module is at Week 26. The last study assessment is at Week 28 for both groups. The end-of-study (EoS) visit for the interchangeability (IC) part of study is planned at Week 28 (ie, 2 weeks after the last study treatment administration, EoS IC).

Extension Phase:

At Week 28, after the EoS IC visit, responsive patients (PASI ≥ 50 [PASI50]) will be offered to continue with the optional open-label Extension Phase (Weeks 28 to 52). AVT02 40 mg will be administered every other week starting from Week 28 (after completing EoS IC assessments), ending with the final study drug administration at Week 50. The EoS visit is planned for Week 52.

The clinical study report (CSR) for the IC part of the study will include the data from the OpenLabel Lead-In Period and Double-Blind Switching Module.

The Extension Phase CSR will include the data from the additional 24-week Open-Label Extension Phase (Weeks 28 to 52).

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed the informed consent form and documentation as required by relevant competent authorities and is able to understand and adhere to the visit schedule and study requirements.
2. Patient is male or female aged 18 to 75 years, inclusive, at the time of Screening.
3. Patients with moderate-to-severe chronic plaque psoriasis who has involved body surface area (BSA) ≥ 10% (Palm Method), ≥ 12 on the PASI, and static Physicians Global Assessments (sPGA) ≥ 3 (moderate) at Screening and at Baseline (Week 1/Day 1).
4. Patient has had stable disease for at least 2 months (ie, without significant changes as defined by the Investigator or designee).
5. Patients with moderate to severe chronic plaque psoriasis who are candidates for systemic therapy or phototherapy, and when other systemic therapies are medically less appropriate.
6. Patient is naive to adalimumab therapy, approved or investigational.
7. Patient has a negative QuantiFERON test for tuberculosis (TB) during Screening. Note: Patients with an indeterminate QuantiFERON test are allowed if they have all of the following:

   1. No evidence of active TB on chest radiograph within 3 months prior to the first dose of study drug.
   2. Documented history of treatment of TB or adequate prophylaxis initiation with an isoniazid-based regimen > 1 month prior to receiving study drug in accordance with local recommendations.
   3. No known exposure to active TB after most recent prophylaxis.
   4. Asymptomatic at Screening and Baseline. Investigators should check with the medical monitor before enrolling such subjects.
8. Women of childbearing potential (except those who are postmenopausal for more than 2 years or if surgically sterile) must have a negative serum pregnancy test during Screening and negative urine pregnancy test at Baseline (Week 1/Day 1).
9. Sexually active women of childbearing potential must agree to use highly effective contraception (sterilization, hormonal contraception pills or injection or implants, sterilization and abstinence) for the duration of the study and until 6 months after the last dose of the study drug. Male patients must agree to use contraception for the duration of the study and agree not to donate sperm during and for 6 months after the last dose of study drug.

Exclusion Criteria:

1. Patient diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, other skin conditions (eg, eczema), or other systemic autoimmune disorder inflammatory disease at the time of the Screening visit that would interfere with evaluations of the effect of the study treatment of psoriasis.
2. Patient has prior use of any of the following medications within specified time periods or will require use during the study:

   1. Topical medications within 2 weeks of Baseline (Week 1/Day 1). PUVA phototherapy and/or UVB phototherapy within 4 weeks prior to the Baseline (Week 1/Day 1).
   2. Nonbiologic psoriasis systemic therapies (eg, cyclosporine, methotrexate, and acitretin) within 4 weeks prior to the Baseline (Week 1/Day 1).
   3. Any prior or concomitant adalimumab therapy, either approved or investigational.
   4. Any systemic steroid in the 4 weeks prior to Screening.
   5. Investigational agent(s) within 90 days or 5 half-lives (whichever is longer) before Baseline (Week 1/Day 1) (Refer to the following table for approved/marketed products).

   Specified washout periods are as follows:
   * Adalimumab: not allowed
   * Alefacept, Briakinumab, Brodalumab, Golimumab: 24 weeks
   * Ustekinumab: 15 weeks
   * Etanercept , Secukinumab , Infliximab , Certolizumab, Pegol: 12 weeks
   * Cyclosporine: 4 weeks
   * Methotrexate: 4 weeks
   * PUVA-UVA/UVB: 4 weeks
   * Oral retinoid: 4 weeks
   * Corticosteroids IM - IV - oral - intra-articular for psoriatic arthritis: 4 weeks
   * Topical psoriasis treatments (except in face, eyes, scalp, palms, soles, and genital area and except only mild potency steroids in these areas): 2 weeks
3. Patient has received live or attenuated vaccines during the 4 weeks prior to Screening or intends to receive a live or attenuated vaccine at any time during the study.
4. Patient has an underlying condition (including, but not limited to, metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious, or gastrointestinal) which, in the opinion of the Investigator or designee, significantly immunocompromises the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy.
5. Patient has a planned surgical intervention during the duration of the study and which, in the opinion of the Investigator or designee, will put the subject at further risk or hinder the patient's ability to maintain compliance with study treatment and the visit schedule.
6. Has any active and serious infection or history of infections as follows:

   1. Any active infection:

      * For which non-systemic anti-infective were used within 4 weeks prior to randomization. Note: patients receiving topical antibiotics for facial acne do not need to be excluded.
      * Which required hospitalization or systemic anti-infective within 8 weeks prior to randomization.
   2. Recurrent or chronic infections or other active infection that, in the opinion of the Investigator or designee, might cause this study to be detrimental to the subject.
   3. Invasive fungal infection or mycobacterial infection.
   4. Opportunistic infections, such as listeriosis, legionellosis, or pneumocystis.
7. Patient is positive for human immunodeficiency virus, hepatitis C virus antibody, or hepatitis B surface antigen (HBsAg) and/or is positive for hepatitis B core antibody.
8. Patient has severe progressive or uncontrolled, clinically significant disease that in the judgment of the Investigator or designee renders the subject unsuitable for the study.
9. Patient has a history of malignancy within 5 years except for adequately treated cutaneous squamous or basal cell carcinoma, in situ cervical cancer, or in situ breast ductal carcinoma.
10. Patient has an active neurological disease, such as multiple sclerosis, Guillain-Barré syndrome, optic neuritis, and transverse myelitis, or a history of neurologic symptoms suggestive of central nervous system demyelinating disease.
11. Patient has moderate to severe heart failure (New York Heart Association [NYHA] Class III/IV).
12. Patient has a history of hypersensitivity to the active substance or to any of the excipients of Humira or AVT02.
13. Patient is pregnant or nursing (lactating) woman, where pregnancy is defined as the state of a female after conception and until the termination of gestation.
14. Patient exhibits evidence (as assessed by the Investigator or designee using good clinical judgment) of active substance abuse (alcohol or drugs) within 6 months of Screening that may impact patient's ability to participate in the study.
15. Is unable to follow study instructions and comply with the protocol in the opinion of the Investigator or designee.
16. Patient has a history of clinically significant hematological abnormalities, including cytopenias (eg, thrombocytopenia, leukopenia).
17. Has a laboratory abnormality that, in the opinion of the Investigator or designee, could cause this study to be detrimental to the subject. The following laboratory abnormalities should be carefully considered:

    1. Hemoglobin < 9 g/dL.
    2. Platelet count < 100,000/mm3.
    3. White blood cell count < 3000 cells/mm3.
    4. Aspartate aminotransferase and/or alanine aminotransferase that is persistently ≥ 2.5 × the upper limit of normal. (Persistently indicates at least on 2 occasions separated by a number of days).
    5. Creatinine clearance < 50 mL/min (Cockcroft-Gault formula).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve over the dosing interval from Week 26 to Week 28 (AUCtau,26-28) | Week 26 to Week 28
  Venous blood samples will be collected for measurement of Area under the plasma concentration-time curve (AUCtau, 26-28) of AVT02 and Humira
Maximum concentration over the dosing interval from Week 26 to Week 28 (Cmax, 26-28) | Week 26 to Week 28
  Venous blood samples will be collected for measurement of serum concentration of AVT02 and Humira

SECONDARY OUTCOMES:
Psoriasis Area and severity index | Week 1 to Week 28 and week 12 to Week 28
  Percent (%) improvement of PASI from Week 1 to Week 28 and from Week 12 to Week 28

CONTACTS AND LOCATIONS:
Overall Officials: Steven Feldman, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (25):
- Georgia (4):
  - 9901, Tbilisi
  - Alvotech Swiss AG - 9904, Tbilisi
  - Alvotech Swiss AG - Site 9902, Tbilisi
  - Alvotech Swiss AG - Site 9903, Tbilisi
- Alvotech Swiss AG - Site 3501, Reykjavik, Iceland
- Poland (7):
  - Alvotech Swiss AG - Site 4803, Gdansk
  - Alvotech Swiss AG - Site 4804, Krakow
  - Alvotech Swiss AG - Site 4807, Krakow
  - Alvotech Swiss AG - Site 4805, Lodz
  - Alvotech Swiss AG - Site 4806, Torun
  - Wromedica Centrum Zdrowia, Wroclaw
  - Alvotech Swiss AG - 4808, Wroclaw
- Russia (6):
  - Alvotech Swiss AG - Site 7001, Kemerovo
  - Alvotech Swiss AG - Site 7005, Krasnodar
  - Alvotech Swiss AG - Site 7003, Saint Petersburg
  - Alvotech Swiss AG - Site 7004, Saint Petersburg
  - Alvotech Swiss AG - Site 7006, Saint Petersburg
  - Alvotech Swiss AG - Site 7002, Saratov
- Ukraine (7):
  - Alvotech Swiss AG - Site 3805, Kharkiv
  - Alvotech Swiss AG - Site 3807, Kharkiv
  - Alvotech Swiss AG - Site 3801, Kyiv
  - Alvotech Swiss AG - Site 3806, Kyiv
  - Alvotech Swiss Ag - Site 3802, Rivne
  - Alvotech Swiss AG - Site 3804, Uzhhorod
  - Alvotech Swiss AG - Site 3803, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feldman SR, Kay R, Reznichenko N, Sobierska J, Dias R, Otto H, Haliduola HN, Sattar A, Ruffieux R, Stroissnig H, Berti F. Assessing the Interchangeability of AVT02 and Humira(R) in Participants with Moderate-to-Severe Chronic Plaque Psoriasis: Pharmacokinetics, Efficacy, Safety, and Immunogenicity Results from a Multicenter, Double-Blind, Randomized, Parallel-Group Study. BioDrugs. 2023 Jul;37(4):551-567. doi: 10.1007/s40259-023-00600-x. Epub 2023 May 19. PMID 37204631